CLINICAL TRIAL: NCT03982875
Title: Efficacy and Application of the Alfred SmartBag System After Ileostomy Creation in Colorectal Surgery: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 11 Heath and Technologies Limited (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11HCCF
Record Dates: First submitted 2019-06-01; First posted 2019-06-12 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Ileostomy - Stoma; Ileostomy; Complications
Keywords: remote monitoring; digital health; ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SmartBag arm (Experimental): The Alfred SmartBag System will be placed on the ostomy site during surgery. The system will be used to wirelessly monitor ostomy function in the hospital setting and the patient will otherwise receive the standard of care. At discharge the patient will continue to use the Alfred SmartBag System and ostomy function will be monitored by the research and clinical teams remotely.
  If participant's output is (i) less than 50mL or greater than 1500mL per day or (ii) greater than 1200mL in two days; the mobile app will alert not only the participant but also the clinical staff (nurse).
  Participants will also receive support from a 'Patient Coach', a trained health coach who is also an ostomy patient to provide quality of life support.
  Interventions: Device: Alfred SmartBag

INTERVENTIONS:
Device: Alfred SmartBag — The Alfred SmartBag encompasses a pouch, a baseplate, and a hub, is intended to be used as a continuous ostomy monitoring system by tracking the volumetric filling of the pouch through integrated thermistor and capacitive sensors and potential leakage and skin irritation development through integrated thermistors in the wafer. The Alfred SmartBag system is indicated for daily use for both in-patient and out-patient settings to provide information to patient and medical professionals. The data is intended to aid patient self-management and to alert the clinical team to changes in the patient condition that may warrant specific intervention.

SUMMARY:
In this study 100 patients due to undergo surgery that will result in an ostomy will be provided with the Alfred SmartBag system. The system encompasses a pouch, a baseplate that can track the volumetric filling of the pouch through integrated thermistor and capacitive sensors and potential leakage and skin irritation development through integrated thermistors in the wafer.

While patients with ileostomy have a risk of dehydration, early identification of those at greater risk may lead to home intervention and decreasing hospital readmission. Decreased readmissions ultimately leads to faster post-operative recovery, decreased risk of complications associated with readmissions (e.i. nosocomial infection, pneumonia, etc.) and decreased healthcare costs. Also evaluating the patients for possible stoma related complications in real time will help in treating them in a timely manner.

DETAILED DESCRIPTION:
Sample size The number of subjects planned to enroll in the study is 100. It is plan to enroll 4 participants per month. Participants will be part of the study from the date of consent to the date when complete the follow-up at 90 days post-surgery.

Selection and screening of potential participants Patients scheduled for office visit with staff physician who will be undergoing to colorectal surgery with new ileostomy creation at the Cleveland Clinic, Main Campus.

Withdraws:

* Participants have the right to withdraw from the study at any time. Written request should be made to the Principal Investigator (PI) via mail. Emre Gorgun, MD, 9500 Euclid Ave. - A30. Cleveland, Oh. 44195
* Participants will be withdrawn from the study if become pregnant.
* Participants will be withdrawn from the study if any type of electronic implants is applied (i.e. pacemakers).
* Participant will be withdrawn per PI and/or sponsor request in the best interest of the participant (e.i. medical condition, technical problems with device or mobile app).
* Before withdrawn, participants will have the opportunity to contact nurse (care coordinator) to request information about changing Alfred SmartBag to regular ostomy bag at their own expense.

Research team:

Principal investigator, co-investigators, research coordinator, nurse (care coordinator), sponsor's representative must be part of the study in IRB and must be compliant with research policies. In addition, everyone in the team must complete CITI and HIPAA in Human Subject Research training courses before engaging in any research activity. No one can take active role in the study without previous documentation and approval by IRB.

Participant enrollment During the preoperative period (average time within 30 days prior to the surgery), eligible patients will be invited to participate in the study by the clinical staff. First, staff physician or clinical personnel will introduce the study. If a patient is interested, the Research Coordinator will explain the study in detail, answer any questions, and provide the informed consent in a quiet clinical setting. If a patient agrees to participate, he/she will sign the informed consent.

Study procedures:

1. Before surgery/introductory session: after signing the informed consent and within 30 days prior to surgery, a participant will meet with the Research Coordinator and sponsor's representative who is certified vendor at Cleveland Clinic, Main Campus. Together, they will provide an extensive training on the Alfred SmartBag system including the ostomy bag and the mobile application. Also, they will assist to set-up the mobile app in the participant's smart phone (e.i. iPhone, Android). This system will allow participant and research study personnel to monitor stoma output daily and in real time. At his time, participant will receive the Alfred Jr. Teddy Bear toy as a part of the "Patient Engagement Program."
2. During the surgery: staff physician will apply the Alfred SmartBag on the ostomy site.
3. Perioperative period (hospitalization/inpatient period): participant will receive standard of care post-operative evaluation and assessment by attending physician and clinical staff. Patient Coaches and certified vendor will contact participant to offer support and answer any question regarding the Alfred Smart Bag system (ostomy bag and mobile app).
4. At discharge from hospital: at the moment of discharge, the participant will receive 30 days-Supply Kit box (complete description of the items can be found on Appendix 2; table 1(p. 29). Participant will be able to monitor ostomy output in real time and contact clinic staff personnel if alerted by the mobile app. In addition, Starbucks gift card $15 dollars and Amazon gift card $25 dollars will be provided.
5. At day 30 post-surgery: second formal wound review will be performed as a part of the standard of care. Documentation of the 30 Day Post-Operative Report. Appendix 2; table 2 (p. 31-34).
6. At day 60 post-surgery: record output in the mobile application. Documentation of the 60 Day Post-Operative Report. Appendix 2; table 2 (p. 31-34).
7. At day 90 post-surgery and beyond: record last output in the mobile app. Documentation of the 90 Day Post-Operative Report. Appendix 2; table 2 (p. 31-34). This is the end of the participation of the study. After this event, participants will not be provided with any part of the Alfred Smart Bag system either ostomy bags, mobile application, or any other services provided as a part of this study. At this time, participants will have the opportunity to choose what type of ostomy bag they prefer to continue with at their own expense.

At any time, complications, unanticipated problems, adverse effects, phone calls, 30-day post-operative report will be documented in logs according to standard practices or in formats included in Appendix 2; table 2 (p.30-31).

ELIGIBILITY:
Inclusion Criteria:

* Older than 22 years of age.
* Ability to communicate in spoken and written English.
* Ability to provide informed consent.
* Scheduled for colorectal surgery with creation of new ileostomy.
* Access to smartphone with bluetooth technology to support mobile and web application.

Exclusion Criteria:

* Pregnancy. Pregnancy test, standard of care, prior to surgery will be reviewed.
* Wearing electronic implants such as pacemakers.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospital readmission within 30 days of surgery | 30 days
  Unplanned hospital readmission will be determined from the hospital patient record. This will be checked by the research team on the 30th postoperative day.

SECONDARY OUTCOMES:
Unplanned hospital readmission within 60 and 90 days of surgery | 60 and 90 days
  Unplanned hospital readmission will be determined from the hospital patient record. This will be checked by the research team on the 60th and 90th postoperative day.
The incidence of high or low output stoma (output <50ml for 1 day, output >1500ml for 1 day or for >1200ml for 2 consecutive days within 30, 60 and 90 days of surgery | 30, 60 and 90 days
  The incidence of high or low output stoma will be determined from the Alfred SmartBag dashboard. A historical report will be analysed at 30, 60 and 90 days.
Number of clinically significant dehydration events within 30, 60 and 90 days of surgery | 30, 60 and 90 days
  Clinically significant dehydration events will be determined from the hospital patient record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.
Emergency department visits within 30, 60 and 90 days of surgery | 30, 60 and 90 days
  Emergency department visits will be determined from the hospital patient record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.
Hydration Clinic visits within 30, 60 and 90 days of surgery | 30, 60 and 90 days
  Hydration clinic visits will be determined from the hospital patient record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.
Surgical Site Infection rates within 30, 60 and 90 days of surgery | 30, 60 and 90 days
  Surgical Site Infection will be determined from the hospital patient record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.
The incidence of patient-reported stoma accidents (leakage) within 30, 60 and 90 days of surgery | 30, 60 and 90 days
  The incidence of patient-reported stoma accidents (leakage) will be determined by analysis of the Patient Coach record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.
Patient reported satisfaction when using the Alfred SmartBag System | 30, 60 and 90 days
  Patient reported satisfaction will be determined by thematic analysis of the Patient Coach record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.
Patient reported quality of life when using the Alfred SmartBag System | 30, 60 and 90 days
  Patient reported quality of life will be determined by thematic analysis of the Patient Coach record. This will be checked by the research team on the 30th, 60th and 90th postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Gorgun, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Department of Colorectal Surgery, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No